CLINICAL TRIAL: NCT01820143
Title: A Phase 1, Randomized, Open-Label, Four-Period Crossover, Multiple-Dose, Single-Center Study to Evaluate the Pharmacokinetics, Pharmacodynamics and Safety Following Administration of Oral Doses of 10, 20 and 40 mg of Ilaprazole and 40 mg of Esomeprazole in Healthy Subjects
Brief Title: Study to Evaluate the Pharmacokinetics, Pharmacodynamics and Safety
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Il-Yang Pharm. Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None
Other Study IDs: Z-P104-099
Record Dates: First submitted 2013-03-25; First posted 2013-03-28 (Estimated); Last update posted 2013-03-28 (Estimated); Status verified 2005-06

CONDITIONS: Healthy; Pharmacokinetics; Pharmacodynamics; Ilaprazole
MeSH Terms: interventions — ilaprazole; Esomeprazole

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (4):
- Treatment sequence ADBC (Experimental): Regimen A: 10 mg of ilaprazole administered QD for 5 days with 240 mL of water. Regimen B: 20 mg of ilaprazole administered QD for 5 days with 240 mL of water. Regimen C: 40 mg of ilaprazole administered QD for 5 days with 240 mL of water. Regimen D: 40 mg of esomeprazole administered QD for 5 days with 240 mL of water.
  Interventions: Drug: Ilaprazole; Drug: Esomeprazole
- Treatment sequence BACD (Experimental): Regimen A: 10 mg of ilaprazole administered QD for 5 days with 240 mL of water. Regimen B: 20 mg of ilaprazole administered QD for 5 days with 240 mL of water. Regimen C: 40 mg of ilaprazole administered QD for 5 days with 240 mL of water. Regimen D: 40 mg of esomeprazole administered QD for 5 days with 240 mL of water.
  Interventions: Drug: Ilaprazole; Drug: Esomeprazole
- Treatment sequence CBDA (Experimental): Regimen A: 10 mg of ilaprazole administered QD for 5 days with 240 mL of water. Regimen B: 20 mg of ilaprazole administered QD for 5 days with 240 mL of water. Regimen C: 40 mg of ilaprazole administered QD for 5 days with 240 mL of water. Regimen D: 40 mg of esomeprazole administered QD for 5 days with 240 mL of water.
  Interventions: Drug: Ilaprazole; Drug: Esomeprazole
- Treatment sequence DCAB (Experimental): Regimen A: 10 mg of ilaprazole administered QD for 5 days with 240 mL of water. Regimen B: 20 mg of ilaprazole administered QD for 5 days with 240 mL of water. Regimen C: 40 mg of ilaprazole administered QD for 5 days with 240 mL of water. Regimen D: 40 mg of esomeprazole administered QD for 5 days with 240 mL of water.
  Interventions: Drug: Ilaprazole; Drug: Esomeprazole

INTERVENTIONS:
Drug: Ilaprazole
Drug: Esomeprazole

SUMMARY:
The objectives of this study were (a) to evaluate the pharmacokinetics and to evaluate and compare the pharmacodynamics of ilaprazole and esomeprazole following a single dose (Day 1) and once daily (QD) administration for 5 consecutive days each of 10-mg, 20-mg, and 40-mg ilaprazole tablets and 40-mg esomeprazole tablets; (b) to evaluate the safety of 10-mg, 20-mg, and 40-mg ilaprazole tablets following QD oral administration for 5 consecutive days; and (c) to characterize the plasma gastrin concentration profile on Day 1 and Day 5 following QD oral administration of 10-mg, 20-mg, and 40-mg ilaprazole and 40-mg esomeprazole tablets for 5 consecutive days.

ELIGIBILITY:
Inclusion Criteria:

* Prior to any study-specific procedures being performed, the subject voluntarily signed the approved informed consent/PIPEDA authorization form after having it fully explained and all questions answered.
* The subject was between 18 and 55 years, inclusive, and was generally in good health.
* Pregnancy test results for all females were negative in order to enter and remain in the study. A serum pregnancy test was performed on all females at Screening, Day -1 of each period, and Day 6 of Period 4 only, or if a subject prematurely discontinued. Results must have been negative in order for study drug to be administered.
* Female subject was using, and agreed to continue the use of, a double-barrier method of birth control. Oral, patch, implants, or injectable contraceptives were accepted as 1 method if the subject had been taking them for greater than 2 months at the Screening Visit. Subjects who had a bilateral tubal ligation, hysterectomy, or bilateral oophorectomy for a minimum of 6 months, or surgical sterilization of partner (vasectomy for 6 months minimum), or were postmenopausal (defined as the absence of menses for 2 years or the absence of menses for 12 months and follicle-stimulating hormone [FSH] level of >40 IU/L) did not require the use of birth control.
* Subject had a negative breath test result for H pylori prior to enrollment.
* At the Screening Visit, subject had a body mass index (BMI) within the range of 18 to 30 kg/m2, as determined by the following calculation.
* Subject was in general good health as evidenced by a medical history, a complete physical examination, and ECG without clinically significant abnormalities.

Exclusion Criteria:

* Subject had current evidence of cardiovascular, central nervous system, hepatic, hematopoietic, renal, or metabolic dysfunction; serious allergy, asthma, history of significant sensitivity to any drug; or lactose intolerance that would contraindicate taking ilaprazole or esomeprazole or would interfere with the conduct of the study.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 40 (Actual)
Dates: Start 2005-02; Primary Completion 2005-04 (Actual); Study Completion 2005-04 (Actual)

PRIMARY OUTCOMES:
Pharmacodynamics of mean pH and percentage of time pH | for 24 hours dosing of Ilaprazole
  For each regimen and day, mean pH and percentage of time pH exceeded 3, 4, 5, and 6 were tabulated and descriptive statistics were provided for 24-hour postdose intervals and each of the following intervals of time relative to dosing: 0 to 4 hours, >4 to 9 hours, >9 to 12 hours, >12 to 16 hours, and >16 to 24 hours.

SECONDARY OUTCOMES:
ilaprazole and esomeprazole plasma concentration data and pharmacokinetic parameter estimates were tabulated and descriptive statistics computed | for 24 hours dosing of Ilaprazole
  The assessments of dose proportionality for ilaprazole regimens were performed via 90% confidence intervals for the ratio of the central values obtained within the framework of the ANOVA on natural logarithms of dose-normalized Cmax, AUCt, and AUC

CONTACTS AND LOCATIONS:
Overall Officials: Gaetano Morelli, MD, Principal Investigator — MDS Pharma Services
Locations (1):
- MDS Pharma Services, Québec, Canada